CLINICAL TRIAL: NCT01356641
Title: Antibiotic Treatment Alone for Acute Simple Appendicitis in Children; a Prospective Cohort Study Part of the Antibiotic Versus Primary Appendectomy in Children (APAC) Trial
Brief Title: Antibiotic Treatment Alone for Acute Simple Appendicitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramon R. Gorter (Other)
Collaborators: Red Cross Hospital Beverwijk (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); St. Antonius Hospital (Other); Flevoziekenhuis (Other)
Responsible Party: Sponsor-Investigator, Ramon R. Gorter, MD, PhD candidate, VU University of Amsterdam
Organization: VU University of Amsterdam (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCA2011/APAC
Record Dates: First submitted 2011-04-18; First posted 2011-05-19 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Appendicitis
Keywords: Antibiotic treatment; Non perforated appendicitis; Children
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic treatment alone (Experimental): Intravenous administration:
  Amoxicillin/clavulanic acid 100/10 mg/kg 6-hourly Gentamicin 7mg/kg once daily
  Oral administration of:
  Amoxicillin/clavulanic acid 50/12.5 mg/kg/day (in three doses)
  Interventions: Drug: Antibiotic treatment alone
- Appendectomy (Active Comparator): Routine appendectomy either laparoscopic or open depending on the surgeon's preference
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Drug: Antibiotic treatment alone — Amoxicillin/clavulanic acid 100/10 mg/kg 6-hourly Gentamicin 7 mg/kg once daily At least 48 hours intravenous administration, in total seven days of antibiotics Oral amoxicillin/clavulanic acid 50/12.5mg/kg
  Arms: Antibiotic treatment alone
Procedure: Appendectomy — Appendectomy either open or laparoscopic depending on the surgeon's preference
  Arms: Appendectomy

SUMMARY:
Appendectomy for acute appendicitis has recently been questioned as being the only correct treatment for appendicitis. Appendectomy has been reported to have significant early and late morbidity. This can be avoided with antibiotic treatment alone. Moreover, better quality of life and lower costs have been associated with antibiotic treatment alone. Five clinical trials in selected patients (males, older than 18 years) comparing appendectomy and antibiotic treatment alone as primary mode of treatment found that antibiotic treatment alone is safe and effective in 48-95% of the patients Conclusive evidence with regard to the efficacy of antibiotic treatment alone in children with proven acute appendicitis however is lacking. We propose a prospective cohort study to answer the following questions:

DETAILED DESCRIPTION:
Primary Objective:

What is the complication rate of the initial antibiotic treatment strategy (IATS) for acute simple appendicitis (radiological proven) in children aged 7-17 years old?

Secondary Objective:

What is the complication rate of the direct appendectomy treatment strategy (DATS) for acute simple appendicitis (radiological proven) in children aged 7-17 years old?

Study design:

Prospective multi-centre pilot cohort study.

Study population:

Children (7-17years old) with radiologically proven simple appendicitis.

Intervention:

Initial antibiotic treatment strategy (IATS): Intravenous administration of amoxicillin/clavulanic acid 25/2.5mg 6-hourly (total 100/10 mg/kg daily; maximum 6000/600mg a day) and gentamicin 7mg/kg once daily will be given for 48 hours. If possible the antibiotics will be switched to oral amoxicillin/clavulanic acid 50/12.5 mg/kg 8-hourly (max 1500/375mg a day) for in total 7 days. If after 72 hours, the patient does not meet the predefined criteria, an appendectomy will be performed.

Control group:

The control group will consist of patients, who do not want the antibiotic treatment. Their medical files will be monitored prospectively. In addition they will be scheduled for an extra outpatient clinic follow up (8 weeks after discharge), extra telephone contact one year after discharge and asked to fill out quality of life questionnaires.

Primary parameters/endpoints:

Safety of initial antibiotic treatment defined as:

Occurrence of major complications, such as:

A. Anaphylactic shock and other allergic reaction to antibiotics administered b. Recurrent appendicitis within 8 weeks c. Recurrent appendicitis within one year after discharge d. Development of perforated appendicitis e. Occurrence of major complaints after delayed appendectomy such as intra-abdominal abscess (IAA), stumpleakage, superficial site infection (SSI), anaesthesia related complications, secondary bowel obstruction (SBO), re-admission, need for re-intervention f. Re-admission g. Re-intervention other than delayed appendectomy

Secondary outcome parameters Major complications associated with appendectomy

1. Stumpleakage
2. Intra-abdominal abscess (IAA)
3. Secondary bowel obstruction (SBO)
4. Superficial site infection (SSI)
5. Need for secondary operation
6. Need for other re-intervention
7. Re-admission
8. Anaesthesia related complication
9. Pneumonia

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

1. Risks of participation: Need for delayed operation, recurrent appendicitis. Risks that are also present in case of non-participation: Allergic reaction to antibiotics, known appendectomy associated complications.
2. Burden of participation: Extra admission day (in comparison with appendectomy), ultrasonography after 48 hours (extra procedure), outpatient follow up (two extra visits), filling out QOL questionnaires. Burden also present in case of non-participation: Intravenous access (normal procedure), daily blood samples (normal procedure). Regarding the control group, the burden will consist of an extra outpatient clinic follow up (8 weeks after discharge), extra telephone contact one year after discharge and fill out quality of life questionnaires.
3. Benefit of participation: Avoidance of surgery and its related early and late morbidity, potential better quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7-17 years
2. Radiologically confirmed simple appendicitis, defined as:

   a. Clinical findings: i. Unwell, but not generally ill ii. Localized tenderness in the right iliac fossa region iii. Normal/hyperactive bowel sounds iv. No guarding v. No mass palpable b. Ultrasonography: i. Incompressible appendix with an outer diameter of ≥6 mm ii. Hyperaemia within the appendiceal wall iii. Without fecalith iv. Infiltration of surrounding fat v. No signs of perforation vi. No signs of intra abdominal abscess/phlegmon

Exclusion criteria:

1. Patients with severe general illness at time of presentation:

   1. Generalized peritonitis defined as:

      Diffuse inflammation of the peritoneum with clinical signs consisting of increasing abdominal pain, generalized tenderness, diffuse abdominal rigidity, sinus tachycardia, signs of paralytic ileus
   2. Severe sepsis or septic shock, as defined by the international paediatric sepsis consensus conference [39]. See attachment 1.
   3. Signs of complex appendicitis
2. Children with a fecalith on ultrasonography.
3. Patients with serious associated conditions or malformations such as:

   1. Congenital or acquired cardiac or pulmonary disease with significant hemodynamic consequences
   2. Immunodeficiency
   3. Malignancy
   4. Homozygous sickle cell disease
   5. Metabolic disorders
4. Patient with documented type 1 allergy to the antibiotics used

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Safety of initial antibiotic treatment strategy | 0-12 months
  Occurrence of major complications, such as:
  A. Anaphylactic shock and other allergic reaction to antibiotics administered b. Recurrent appendicitis within 8 weeks c. Recurrent appendicitis within one year after discharge d. Development of perforated appendicitis e. Occurrence of major complaints after delayed appendectomy such as intra-abdominal abscess (IAA), stumpleakage, superficial site infection (SSI), anaesthesia related complications, secondary bowel obstruction (SBO), re-admission, need for re-intervention f. Re-admission g. Re-intervention other than delayed appendectomy

SECONDARY OUTCOMES:
Safety of the direct appendectomy treatment strategy | 0-12 months
  Major complications associated with appendectomy
  1. Stumpleakage
  2. Intra-abdominal abscess (IAA)
  3. Secondary bowel obstruction (SBO)
  4. Superficial site infection (SSI)
  5. Need for secondary operation
  6. Need for other re-intervention
  7. Re-admission
  8. Anaesthesia related complication
  9. Pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Ramon R Gorter, MD, Principal Investigator — Amsterdam UMC, location VUmc; Hugo A Heij, MD, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (4):
- Netherlands (4):
  - Flevoziekenhuis, Almere Stad
  - Academic medical center of Amsterdam, Amsterdam
  - VU University medical center, Amsterdam
  - Red Cross Hospital, Beverwijk